CLINICAL TRIAL: NCT01308957
Title: Omega-3 Fatty Acids, Muscle Mass and Muscle Function
Brief Title: Fish Oil and Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201012999
Record Dates: First submitted 2011-02-25; First posted 2011-03-04 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Fatty Acids, Omega-3; Omacor; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Long chain omega-3 fatty acids (Experimental)
  Interventions: Dietary Supplement: Omega-3 fatty acids
- Corn oil (Placebo Comparator)
  Interventions: Dietary Supplement: corn oil
- Young healthy controls (No Intervention): Young subjects' muscle mass and physical function will be evaluated once (i.e., during baseline testing only). The data in young subjects will be used to determine the magnitude of the aging-induced decline in muscle mass and physical function in the older subjects prior to starting the interventions.

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — 4 grams per day for 24 weeks
  Other Names: Lovaza
  Arms: Long chain omega-3 fatty acids
Dietary Supplement: corn oil — 4 grams per day for 24 weeks
  Arms: Corn oil

SUMMARY:
The purpose of this study is to examine the effect of omega-3 fatty acid supplementation on changes in muscle mass, muscular strength and physical function.

DETAILED DESCRIPTION:
Loss of muscle mass is a normal consequence of aging in many older adults, worsened by chronic illness, poor appetite and diet, and reduced physical activity. The ensuing decline in physical function is a major cause of frailty, disability and death. Treatments that can reverse or reduce the age-associated loss of muscle mass are therefore much needed. Evidence is emerging that consumption of fish or fish oil derived long-chain omega-3 polyunsaturated fatty acids (LCn-3PUFA) may be important for maintenance of muscle mass and physical function throughout the life-span. However, the effect of LCn-3PUFA supplementation on muscle mass, muscle strength and overall physical function is not known. The goal of this study therefore is to determine the effect of LCn-3PUFA supplementation on muscle mass, muscle strength and physical function in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese (i.e., BMI less than 35 kg/m2)
* Between 18 to 45 or between 60 and 85 y old
* Subjects who are sedentary (<1 h of exercise/week)

Exclusion Criteria:

* Subjects with evidence of significant organ system dysfunction (e.g. diabetes, severe cardiovascular disease, hyperlipidemia, cirrhosis, hypogonadism, uncontrolled hypo- or hyperthyroidism; uncontrolled hypertension)
* Subjects with metal implants
* Subjects with iron storage disease,
* Subjects with severe ambulatory impairments,
* Individuals with cancer or cancer that has been in remission for <5 years,
* Individuals with dementia,
* Individuals who smoke,
* Subjects who are taking medications known to affect muscle (e.g., steroids),
* Subjects who receive anticoagulant therapy.
* Subjects taking medications to control certain medical conditions (e.g., hypertension) will be included if the drug regimen has been stable for at least 6 months before entering the study and is not expected to change during the study.
* Subjects with allergies to sea food,
* Subjects who regularly consume fish oil or consume >2 servings of fish with a high LCn-3PUFA content (e.g. salmon, mackerel, sardines, etc) per week.
* Physical performance test score less than 17 out of 36.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of omega-3 fatty acids on muscle mass | Change from baseline in muscle mass at 24 weeks in older adults only
  We will measure thigh muscle volume by using magnetic resonance imaging. These measurements will also be assessed at week 12 in a subset of subjects but the data will not be used as a primary outcome measure.
Evaluate the effect of omega-3 fatty acids on physical function | Change from baseline in physical function at 24 weeks in older adults only
  We will evaluate muscle strength by assessing one-repetition maximum strength of upper- and lower-body skeletal muscles, grip strength and isometric and isokinetic force development. We will assess overall physical function using the physical performance tests, which evaluates the ability to perform usual daily activities such as climbing a flight of stairs, walking 50 feet and putting on and removing a coat. These measurements will also be assessed at week 12 in a subset of subjects but the data will not be used as a primary outcome measure.

SECONDARY OUTCOMES:
Evaluate the effect of aging on muscle mass | During baseline testing in both young and older subjects
  We will measure total fat-free mass by duel X-ray absorptiometry, thigh muscle and intermuscular fat volumes by using magnetic resonance imaging.
Evaluate the effect of aging on physical function | During baseline testing in both young and older subjects
  We will evaluate muscle strength by assessing one-repetition maximum strength of upper- and lower-body skeletal muscles, grip strength, thigh isometric and isokinetic force development and time-to-peak force development during thigh isokinetic exercises. We will assess overall physical function using the physical performance tests, which evaluates the ability to perform usual daily activities such as climbing a flight of stairs, walking 50 feet and putting on and removing a coat.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Smith GI, Julliand S, Reeds DN, Sinacore DR, Klein S, Mittendorfer B. Fish oil-derived n-3 PUFA therapy increases muscle mass and function in healthy older adults. Am J Clin Nutr. 2015 Jul;102(1):115-22. doi: 10.3945/ajcn.114.105833. Epub 2015 May 20. PMID 25994567